CLINICAL TRIAL: NCT06333704
Title: A Multi-Centre, Prospective, Observational Post-Marketing Surveillance to Investigate the Long-Term Safety of SPIKEVAX BIVALENT and SPIKEVAX X Injection Under Routine Clinical Care in Korea
Brief Title: Post-marketing Surveillance (PMS) Use-Result Surveillance With SPIKEVAX BIVALENT and SPIKEVAX X Injection.
Status: Recruiting | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P924
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SPIKEVAX BIVALENT or SPIKEVAX X: Participants receiving at least 1 dose of SPIKEVAX BIVALENT vaccine or SPIKEVAX X Injection are monitored for safety parameters up to 28 days post vaccination.
  Interventions: Biological: SPIKEVAX Bivalent; Biological: SPIKEVAX X

INTERVENTIONS:
Biological: SPIKEVAX Bivalent — No study drug will be administered during this study as this is an observational study.
  Other Names: SPIKEVAX Bivalent BA.1; SPIKEVAX BIVALENT BA.4/5; SARS-CoV-2-mRNA vaccine
Biological: SPIKEVAX X — No study drug will be administered during this study as this is an observational study.
  Other Names: SPIKEVAX XBB.1.5; SARS-CoV-2-mRNA vaccine

SUMMARY:
The main objective of the surveillance is to evaluate the incidence of the adverse events (AEs), and other safety related information in South-Korean population.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be 18 years or older for Spikevax bivalent BA.1, SPIKEVAX BIVALENT BA.4/5 vaccine, and 12 years or older for Spikevax XBB.1.5 injection.
* Participants of any age which is approved for the use of SPIKEVAX BIVALENT BA.1, SPIKEVAX BIVALENT BA.4/5 or SPIKEVAX XBB.1.5 for active immunization to prevent COVID-19 caused by SARS-CoV-2.
* Participant who will be vaccinated with SPIKEVAX BIVALENT BA.1, SPIKEVAX BIVALENT BA.4/5 or SPIKEVAX XBB.1.5 following local label approved by Ministry of Food and Drug Safety (MFDS).
* Participant who will be vaccinated with at least one dose of SPIKEVAX BIVALENT BA.1, SPIKEVAX BIVALENT BA.4/5 or SPIKEVAX XBB.1.5.

Exclusion Criteria:

* Participant whose participation is deemed inappropriate at the investigator's discretion.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey is Korean participants vaccinated with SPIKEVAX BIVALENT or SPIKEVAX X injection who meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 4206 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2028-12-10 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With AEs | Up to 28 days post vaccination

CONTACTS AND LOCATIONS:
Locations (24):
- South Korea (24):
  - Yonseimin Clinic, Wŏnju, Gangwon-do
  - Hyundai Clinic, Bucheon-si, Gyeonggi-do
  - Ma Hak ki Family Medicine Clinic, Bucheon-si, Gyeonggi-do
  - Nalee Hospital, Gimpo-si, Gyeonggi-do
  - COA ENT Clinic, Goyang-si, Gyeonggi-do
  - Joon Pediatric Clinic, Gwangmyeong, Gyeonggi-do
  - Janghyeon Medicine Clinic, Siheung, Gyeonggi-do
  - Hanyang Union Rehabilitation Medicine Clinic, Yangju, Gyeonggi-do
  - KimHyungjoo Clinic, Yangju, Gyeonggi-do
  - Kium Children Hospital, Gunsan, Jeollabuk-do
  - Sinsegie ENT Clinic, Busan
  - Jeil Family Medicine Clinic, Gwangju
  - Bupyeong Yonsei Medical Clinic, Incheon
  - Inha University Hospital, Incheon
  - Woori Medical Clinic, Seoul
  - Yonsei Kids Pediatrics Clinic, Seoul
  - Star Pediatrics Clinic, Seoul
  - Seoul Bon Clinic, Seoul
  - Dr Cho's Family Medical Clinic, Seoul
  - Songpa Korea Neurosurgical Clinic, Seoul
  - GF Pediatrics Clinic, Seoul
  - Kim Il Joong Internal Medicine Clinic, Seoul
  - New Yonsei ENT Clinic, Seoul
  - Soo Orthopedics Clinic, Seoul